CLINICAL TRIAL: NCT02531555
Title: Clinical Efficacy Of 810 Nanometer Diode Laser As An Adjunct To Mechanical Periodontal Treatment Of Residual Periodontal Pockets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Meseli et al.
Record Dates: First submitted 2015-08-06; First posted 2015-08-24 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Periodontitis
Keywords: chronic periodontitis; dental scaling; gingival crevicular fluid; lasers; periodontal pocket; root planing
MeSH Terms: conditions — Chronic Periodontitis; Periodontal Pocket

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group M (Active Comparator): Mechanical periodontal treatment (Group M): Scaling and root planing were performed with Gracey curettes until the operator feels that root surface is clean, hard and smooth.
  Interventions: Device: Gracey curettes
- Group L (Experimental): Pocket disinfection with diode laser (Group L): Subgingival irradiation with a GaAlAs diode laser (CHEESE®, Gigaa Laser, China) was applied to residual pockets each for 20 sec in continious mode. The diode laser had a wavelenght of 810 nm and power output of 1 W for subgingival irradiation (Maximum output power of device was 7 W). Diode laser application was performed parallel to root surface by a 200 µm fiber tip inserted at the bottom of periodontal pocket and slowly moved from apical to coronal direction in a sweeping motion without local anesthesia.
  Interventions: Device: 810 Nanometer Wavelenght GaAlAs Diode Laser
- Group M+L (Experimental): Combined treatment (Group M+L): Following mechanical periodontal treatment, pocket irradiation with diode laser was performed as mentioned above.
  Interventions: Device: 810 Nanometer Wavelenght GaAlAs Diode Laser; Device: Gracey curettes

INTERVENTIONS:
Device: 810 Nanometer Wavelenght GaAlAs Diode Laser — FDA approved 810 nanometer GaAlAs Diode Laser
  Other Names: CHEESE®, Gigaa Laser, China
  Arms: Group L; Group M+L
Device: Gracey curettes
  Other Names: Hu-Friedy, SG 5/6, 7/8, 11/12, 13/14, Hu-Friedy Ins. Co., USA
  Arms: Group M; Group M+L

SUMMARY:
Background: Aim of this randomized controlled parallel-designed study was to evaluate the effects of diode laser as an adjunct to mechanical periodontal treatment on clinical parameters and gingival crevicular fluid (GCF) volume of the residual pockets diagnosed following initial periodontal treatment in chronic periodontitis (CP) patients.

Methods: A total of 84 residual pockets on single-rooted teeth in 11 CP patients were included and randomly assigned into 3 groups. Residual pockets were treated either only by mechanical treatment (Group M) (n=28), only by diode laser disinfection (Group L) (n=28) or by combination of these techniques (Group M+L) (n=28). Plaque index, gingival index (GI), bleeding on probing (BoP), probing depth (PD), clinical attachment level and gingival recession were assessed at baseline and 8 weeks after treatment of residual pockets. GCF samples were collected at baseline, 1 and 8 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy,
* Non-smoker,
* Chronic periodontitis diagnosed according to Armitage 1,
* Aged between 35 and 65,
* Not received any periodontal treatment within the last 3 months,
* Have horizontal bone loss radiographically,
* Presence at least 20 natural teeth except third molars
* Consent to participate in the study.

Exclusion Criteria:

* Any systemic disease that might interfere with the prognosis of periodontal disease (i.e. diabetes mellitus, HIV infection),
* Smoking,
* Antibiotics, anti-inflammatory drugs or any other medication taken within the previous 6 months that may affect the outcome of the study,
* Any physical limitations or restrictions that might preclude normal oral hygiene procedures.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Probing depth | 8 week
  Probing depth is defined as the distance from the free gingival margin to the bottom of the periodontal pocket.

SECONDARY OUTCOMES:
Plaque index | 8 week
Gingival index | 8 week
Clinical attachment level | 8 week
  Clinical attachment level is defined as the distance from the cementoenamel junction to the bottom of the periodontal pocket
Bleeding on probing via periodontal probe | 8 week
  Bleeding on probing is defined as presence of bleeding from gingival sulcus during the probing of this area via periodontal probe.
Change of gingival crevicular fluid volume | Baseline, 8 weeks
  Gingival crevicular fluid is a blood-originated fluid playing important determinanat role in the ecology of the gingival sulcus and periodontal pocket

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Faculty of Dentistry, Istanbul, Turkey (Türkiye)